CLINICAL TRIAL: NCT02530073
Title: Pilot Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in Severe Left Congenital Diaphragmatic Hernia (CDH)
Brief Title: Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) for CDH
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Crombleholme, Director of Fetal Care Center, Connecticut Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-133; NCT06064188 (obsolete NCT alias)
Record Dates: First submitted 2015-07-31; First posted 2015-08-20 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Congenital Diaphragmatic Hernias
Keywords: congenital diaphragmatic hernia; FETO; tracheal occlusion
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fetoscopic Endoluminal Tracheal Occlusion (FETO) (Experimental): An un-blinded non-randomized single arm pilot study of FETO in fetuses with congenital diaphragmatic hernia (CDH)
  Interventions: Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO)

INTERVENTIONS:
Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO) — This study will position and remove an endoluminal tracheal balloon in utero (FETO) to study the feasibility of implementing FETO therapy in the most severe group of fetuses with left CDH and observed/expected length head ratio <25% (O/E LHR).
  Other Names: BALT GOLDBAL2 Tracheal Balloon Catheter system

SUMMARY:
The rationale for fetal therapy in severe congenital diaphragmatic hernia (CDH) is to restore adequate lung growth for neonatal survival.

DETAILED DESCRIPTION:
Prenatal tracheal occlusion (TO) obstructs the normal egress of lung fluid during pulmonary development leading to increased lung tissue stretch, increased cell proliferation, and accelerated lung growth. European colleagues have developed foregut endoscopy and techniques to position and remove endoluminal tracheal balloons in utero. Recently, the Belgium group published summary results of FETO showing an improved survival in 175 patients with isolated left CDH from 24% to 49%.

The goal of this pilot study is to study the feasibility of implementing FETO therapy in the most severe group of fetuses with left CDH Observed/expected lung-to-head ratio < 25%(O/E LHR < 25%).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years and older, who are able to consent
* Singleton pregnancy

Fetal

* Normal Karyotype
* Fetal Diagnosis of Isolated Left CDH with liver up
* Gestation at enrollment prior to 29 wks plus 6 days
* SEVERE pulmonary hypoplasia with Ultra Sound O/E LHR < 25%

Exclusion Criteria:

* Pregnant women <18 years of age.
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* Technical limitations precluding fetoscopic surgery
* Rubber latex allergy
* Preterm labor, cervix shortened (<15 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Psychosocial ineligibility, precluding consent
* Diaphragmatic hernia: right-sided or bilateral, major associated anomalies, isolated left-sided with the O/E LHR ≥ 25%
* Inability to remain at FETO site during time period of tracheal occlusion, delivery and postnatal care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Percent of neonatal survivors at time of discharge | Discharge from the hospital, an expected average of 12 weeks.
  Feasibility, safety, and survival rates of the FETO procedure

SECONDARY OUTCOMES:
Prenatal increase in lung volume | 2 weeks (prenatally)
  Lung volume after FETO procedure
Number of days of Postnatal mechanical ventilator support | First 28 days of postnatal life
  mechanical ventilator support will be monitored and recorded in days of use
Changes in RNA content of tracheal and amniotic fluid | At time of balloon placement and removal
  Describe how tracheal occlusion affects the RNA content of amniotic and tracheal fluid in CDH fetuses, and to correlate this transcriptomic profile to the degree of lung hypoplasia and fetal and neonatal clinical outcomes.
Characterization of extracellular vesicles (EVs) and miRNAs in tracheal and amniotic fluid | At time of balloon placement and removal
  To describe how extracellular vesicles (EVs) are derived from the amniotic and tracheal fluid of CDH patients before and after tracheal occlusion, and to determine whether the identified miRNAs of interest are intra- or extra-vesicular.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Crombleholme, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States